CLINICAL TRIAL: NCT03689166
Title: Effect of Probiotics on the Preterm Delivery Rate (< 37 Weeks) in Pregnant Women at High Risk for Preterm Birth (Pregnant Women With Threatened Preterm Labour): PROPEV TRIAL Protocol
Brief Title: Effect of Probiotics on the Preterm Delivery Rate in Pregnant Women at High Risk for Preterm Birth
Acronym: PROPEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal-Infantil Vall d´Hebron Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR(AMI)236/2016
Record Dates: First submitted 2018-02-11; First posted 2018-09-28 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Preterm Birth
Keywords: Probiotics; Preterm birth; Threatened preterm labour
MeSH Terms: conditions — Premature Birth | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Definition and design. Prospective, double-blind randomised study.
  Population Pregnant women admitted for TPL between weeks 24.0 and 34.6 of gestation at the participating centre.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Active Comparator): Probiotic drug
  Interventions: Dietary Supplement: Probiotic
- Control group (Placebo Comparator): This group will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Reduce preterm birth with this dietary supplement
  Arms: Probiotics group
Other: Placebo — Placebo
  Arms: Control group

SUMMARY:
Preterm birth (PB) continues to be the main cause of perinatal morbidity and mortality, with emotional and economic consequences. Despite improvements in health, PB prevalence remains stable, possibly due to complex causes such as maternal age, stress, multiparity, etc. Shortening of the uterine cervix in early stages of gestation is a risk factor for PB. The presence of abnormal vaginal microbiota in the early stages of pregnancy is als a risk factor for PB. However, no studies have analysed the impact of probiotics (live microorganisms which, in adequate amounts, confer a health benefit on the host) on the PB in high-risk PB patients (pregnant women with threatened preterm delivery, i.e., uterine contractions and cervical shortening, with a 30% PB risk before 34 weeks, and 50% PB prior to 37 weeks (> 6-10% PB). Similarly, the effect of probiotics on vaginal flora dominated by lactic acid-producing bacteria could be analysed.

DETAILED DESCRIPTION:
Hypothesis

* Pregnant women with threatened preterm labour (TPL) will present vaginal microbiome different from those without TPL.
* Treatment with probiotics will modify the vaginal microbioma of pregnant women with TPL.
* The PB rate before 37 weeks in pregnant women with TPL who have received probiotics since their diagnosis will be reduced by at least 30%.

Goals

* To correlate the use of probiotics of pregnant women with TPL with the PB rate before 37 weeks.
* To ascertain the PB rate before 28, 30, 32 and 34 weeks in both groups.
* To assess neonatal morbidity between both groups.

Methods

Prospective, randomised, longitudinal, prospective, double-blind study.

Relevance

This study will determine whether the use of probiotics in pregnant women with TPL is associated with a lower risk of PB before 37 weeks. If so, it would allow us to act on the tertiary prevention of PB and treatment of TPL, the main cause of perinatal morbidity and mortality in our setting. It will also facilitate understanding of the pathophysiology of PB, influence of vaginal microbiota and the mechanism of action of probiotics.

ELIGIBILITY:
Inclusion criteria

* Threatened preterm labour: regular clinical and cardiotography-registered uterine dynamics, and cervical modifications (cervical shortening ≤ 25 mm between 24 and 29 weeks, and ≤ 15 mm between 30 and 34 weeks) according to our care protocol.
* Single gestation.
* Echographically-normal foetal morphology.
* Minimum age 18 years.
* Ability to understand informed consent.
* Signed informed consent.

Exclusion criteria

* Multiple gestations.
* Pregnant women with diagnosis of chorioamnionitis.
* Cervical dilation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Preterm birth rate <37 weeks | From 24 to 37 weeks
  To evaluate the percentage of preterm birth in each group (in days of gestation)

SECONDARY OUTCOMES:
Preterm birth rate <34 weeks | From 24 to 34 weeks
  To evaluate the percentage of preterm birth in each group (in days of gestation)
Preterm birth rate <32 weeks | From 24 to 32 weeks
  To evaluate the percentage of preterm birth in each group (in days of gestation)
Preterm birth rate <30 weeks | From 24 to 30 weeks
  To evaluate the percentage of preterm birth in each group (in days of gestation)
Preterm birth rate <28 weeks | From 24 to 38 weeks
  To evaluate the percentage of preterm birth in each group (in days of gestation)
Intergroup neonatal morbidity | First year of life of newborns
  To assess neonatal morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Herbron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This study will allow us to determine whether the use of probiotics in pregnant women with TPL is associated with an increased risk of PB. If so, it would allow us to act on the tertiary prevention of PB and treatment of TPL, the main cause of perinatal morbidity and mortality in our setting. Similarly, it will facilitate understanding of the pathophysiology of PB, influence of vaginal microbiota and the mechanism of action of probiotics.

REFERENCES:
- [Derived] Del Barco E, Molano LG, Vargas M, Miserachs M, Puerto L, Garrido-Gimenez C, Soler Z, Munoz B, Pratcorona L, Rimbaut S, Vidal M, Dalmau M, Casellas A, Carreras E, Manichanh C, Goya M. The Effect of Probiotics on Preterm Birth Rates in Pregnant Women After a Threatened Preterm Birth Episode (The PROPEV Trial). Biomedicines. 2025 May 8;13(5):1141. doi: 10.3390/biomedicines13051141. PMID 40426968